CLINICAL TRIAL: NCT00752414
Title: Phase 1b, Randomized, Single-Blind, Placebo-Controlled, Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MP-376 Inhalation Solution Administered for 5 Days to Chronic Bronchitis Patients
Brief Title: A Phase 1b Study to Evaluate the Safety and PK of MP-376 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mpex-301
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MP-376 Inhalation Solution
  Interventions: Drug: MP-376 (Levofloxacin solution for Inhalation)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP-376 (Levofloxacin solution for Inhalation) — Daily for 5 days
  Arms: 1
Drug: Placebo — same frequency as MP-376
  Arms: 2

SUMMARY:
Patients with Chronic Obstructive Pulmonary Disease (COPD) suffer from frequent and recurrent acute exacerbations (AECB) which are associated with enormous healthcare expenditures and significant morbidity, specifically an increased risk of death, a decline in pulmonary function and a significant change in quality of life. Bacteria appear to have an important role in acute exacerbations in chronic bronchitis and COPD. Studies of acute exacerbations in COPD have shown a reduction in bacterial load with prolonged exacerbation-free interval. In addition, recent studies indicate that acquisition of a new strain of H. influenzae, M. catarrhalis, S. pneumoniae or P. aeruginosa are responsible for many of these exacerbations. Chronic inflammation and bacterial infection predispose many patients to frequent and recurrent acute exacerbations.

Mpex, (the sponsor on record at time of the study's initial registration) believes that intermittent administration of inhaled MP-376 in high risk patients will decrease the incidence of acute exacerbations by both by lowering the organism burden, and resultant inflammation, as well as pre-emptive eradication of any newly acquired bacterial strains.

DETAILED DESCRIPTION:
This study will be a Phase 1b, multi-center, randomized, single-blind, placebo-controlled study to evaluate the safety, tolerability, and pharmacokinetics of MP-376 solution for inhalation given for 5 days to COPD patients.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* >/= 40 years of age
* History of COPD
* FEV1 </= 65% of predicted and FEV1/FVC </= 0.7 value at Screening
* Clinically stable with no changes in health status within the last 30 days
* Lifetime smoking history of at least 15 pack-years
* Willing and able to give informed consent

Exclusion Criteria (selected):

* Use of any systemic or inhaled antibiotics within 30 days prior to baseline
* History of hypersensitivity to fluoroquinolones or intolerance with aerosol medication
* CrCl < 50/ml/min, AST, ALT or total bilirubin >/= 3 x ULN at Screening
* Significant or unstable medical conditions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability and PK of two dosage regimens of MP-376 | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (5):
- United States (5):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Omaha, Nebraska
  - Buffalo, New York
  - Columbus, Ohio